CLINICAL TRIAL: NCT03979755
Title: Pelvic Floor Dysfunction in Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Aline Moreira Ribeiro, Principal Investigator, University of Sao Paulo
Other Study IDs: 3.358.945
Record Dates: First submitted 2019-06-02; First posted 2019-06-07 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Cancer; Pelvic Floor Dysfunction
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Women cancer survivors living in Campo Belo, Minas Gerais.
  Interventions: Other: Application of questionnaires
- Control Group: Women in routine follow-up in the public health system in Campo Belo, Minas Gerais.
  Interventions: Other: Application of questionnaires

INTERVENTIONS:
Other: Application of questionnaires — Application of questionnaires described by telephone.

SUMMARY:
Introduction: Pelvic floor dysfunctions (PFD) represent a major public health problem manifested through lower urinary tract symptoms (LUTS), anorectal and sexual dysfunction. PFD is a common problem in cancer survivors with a negative impact on quality of life (QoL). However, the magnitude of its prevalence in women with no history of cancer is unknown. Aims: To verify the prevalence of PFD among cancer survivors. Secondly, to evaluate sexual function, QoL and functional performance of women cancer survivors and the influence of PAD on QoL, ADL and emotional health. Methods: Two group is being conducted. Study Grourp (SG) are women diagnosed with any neoplasia in the period between 2013 and 2017 living in the municipality of Campo Belo / MG. Control Group (CG) are women in routine clinical follow-up at the units of the Family Health Program of that city, with no history of cancer. All volunteers will be interviewed by telephone through the application of a structured questionnaire that assesses socioeconomic indicators, gynecological-obstetric history and life habits, as well as specific questionnaires for the evaluation of PFD, functional performance and QoL.

DETAILED DESCRIPTION:
Data collect: The lists of women residing in Campo Belo / MG, with and without a history of cancer, were used by the Municipal Health Department (MDH). Data on cancer treatment may also be used, if they are in the field of MDH. The information used in this study originated in a questionnaire developed for the study that included socioeconomic indicators, gynecological-obstetric history and life habits (smoking, alcohol consumption and sedentary lifestyle). All interviews were conducted by telephone. Other questionnaires were also used, all translated and validated for Brazilian Portuguese.

SG and CG groups were matched for age and parity. Age information was collected continuously and grouped into class intervals from the age of 20, resulting in strata for analysis with cohort points at 20, 30, 40, 50, 60, 70 and 80 years. Parity was divided into five categories according to the parity: nulliparous, 1 delivery, 2 delivery, 3 delivery, 4 or more deliveries.

Variables

Primary variable:

(A) Prevalence of PFD: The Pelvic Floor Disability Index (PFDI-20) was used to evaluate the prevalence and symptomatology of pelvic organ prolapse (POP), anorectal symptoms and urinary incontinence (UI) (Barber et al., 2005; Arouca et al., 2016).

Secondary variables:

(A) Sexual function: The Sexual Questionnaire for Urinary Incontinence and Pelvic Organ Prolapse (PISQ-12) evaluated the sexual function and prevalence of sexual dysfunction in the sample (Rogers et al. , 2003; Santana et al., 2012).

(B) Quality of life: The World Health Organization Quality of Life Questionnaire - Brief (WHOQOL-BREF) (Fleck et al., 2000) was used for the evaluation of QoL.

(C) Functional performance: In order to evaluate the functional performance of the sample (real level of human function, self-care capacity and level of ambulation), the Functionality Assessment Flowchart (FAF) developed by Paiva et al 2015.

(D) Influence of PFD on QoL and AVD: The Pelvic Floor Impact Questionnaire (PFIQ-7) was used to assess the impact of PFD on QoL, ADL and emotional health (Barber et al., 2005; Arouca et al., 2016).

ELIGIBILITY:
Inclusion Criteria:

Study Group:

* Women living in the city of Campo Belo, Minas Gerais who had cancer in the period between 2013 and 2017.

Control Group:

* Women in routine follow-up in the public health network through the units of the Family Health Program of the city of Campo Belo, Minas Gerais, without previous clinical history of cancer.

Exclusion Criteria:

* Women that have more than one tumor;
* Women with metastatic disease;
* Women do not have the physical and mental conditions to respond to the interviews;
* No acceptance or consent to participate in the survey.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study Group: women surviving cancer residing in the municipality of Campo Belo, Minas Gerais, with prior cancer treatment and diagnosis confirmed by histopathology in the last five years (2013-2017).
  Control Group: women in routine follow-up in the public health network through the units of the Family Health Program of the city of Campo Belo, Minas Gerais, with pathologies not associated positively or negatively with the exposures of interest of the study. The controls do not present a present or previous clinical history of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Initial screening | Three months
  Initial screening of the number of women with cancer in the period between 2013 and 2017
Application of questionnaries | Three months
  Application of questionnaries by telephone

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arouca MA, Duarte TB, Lott DA, Magnani PS, Nogueira AA, Rosa-E-Silva JC, Brito LG. Validation and cultural translation for Brazilian Portuguese version of the Pelvic Floor Impact Questionnaire (PFIQ-7) and Pelvic Floor Distress Inventory (PFDI-20). Int Urogynecol J. 2016 Jul;27(7):1097-106. doi: 10.1007/s00192-015-2938-8. Epub 2016 Jan 19. PMID 26782099
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Fitz FF, Santos ACC, Stüpp L, Bernardes APMR, Marx AG. Impacto do tratamento do cancer de colo uterino no assoalho pélvico. FEMINA. 2011;39(8):387-93.
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Background] INTERNATIONAL AGENCY OF RESEARCH ON CANCER. Cancer Incidence in Five Continents, Lyon: IARC Scientific Publications, 1992.
- [Background] Instituto Nacional de Câncer José Alencar Gomes da Silva. Coordenação de Prevenção e Vigilância. Estimativa 2018: incidência de câncer no Brasil / Instituto Nacional de Câncer José Alencar Gomes da Silva. Coordenação de Prevenção e Vigilância. Rio de Janeiro: INCA, 2017.
- [Background] Paiva CE, Siquelli FA, Santos HA, Costa MM, Massaro DR, Lacerda DC, Nunes JS, de Padua Souza C, Paiva BS. The Functionality Assessment Flowchart (FAF): a new simple and reliable method to measure performance status with a high percentage of agreement between observers. BMC Cancer. 2015 Jul 5;15:501. doi: 10.1186/s12885-015-1526-0. PMID 26142726
- [Background] Rogers RG, Coates KW, Kammerer-Doak D, Khalsa S, Qualls C. A short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J Pelvic Floor Dysfunct. 2003 Aug;14(3):164-8; discussion 168. doi: 10.1007/s00192-003-1063-2. Epub 2003 Jul 25. PMID 12955337
- [Background] Santana GW, Aoki T, Auge AP. The Portuguese validation of the short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J. 2012 Jan;23(1):117-21. doi: 10.1007/s00192-011-1505-1. Epub 2011 Jul 28. PMID 21796471